CLINICAL TRIAL: NCT03591692
Title: Comparison of Anterior Cervical Anteriodisplacement Fusion and Corpectomy Decompression Fusion in Treatment of Ossification of the Posterior Longitudinal Ligament: A Multi-center，Controlled, Randomized, Open Label Clinical Study
Brief Title: A Multi-center Study：Comparison of ACAF and ACCF in the Treatment of Cervical OPLL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Xuzhou No.1 Peoples Hospital (Other); Jiangxi Provincial People's Hopital (Other); No.102 Military Hospital of China Dormitory Area (Other); Shanghai Kaiyuan Orthopedic Hospital (Unknown); Huaibei Coal Mine General Hospital (Unknown)
Responsible Party: Principal Investigator, Jiangang Shi, Chief of No.2 department of spinal surgery, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CZ1805OPLL
Record Dates: First submitted 2018-06-06; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Ossification of Posterior Longitudinal Ligament
MeSH Terms: conditions — Ossification of Posterior Longitudinal Ligament

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistical analysist do not know the group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACAF surgery (Experimental): Underwent anterior controllable antedisplacement and fusion
  Interventions: Procedure: ACAF surgery
- ACCF surgery (Placebo Comparator): Underwentanterior controllable antedisplacement and fusion
  Interventions: Procedure: ACCF surgery

INTERVENTIONS:
Procedure: ACAF surgery — The main surgical procedures include discectomy of the involved levels, thinning of the anterior part of the involved vertebrae, intervertebral cages, anterior plate and screws installation, bilateral osteotomies of the vertebrae, and antedisplacement of the vertebrae-OPLL complex
  Arms: ACAF surgery
Procedure: ACCF surgery — Removal of the vertebral body，exposed ossification of the posterior longitudinal ligament，and then removed
  Arms: ACCF surgery

SUMMARY:
Background:The ACAF technology has been in clinical trials for some time. More and more doctors are starting to pay attention to this technology. There are many hospitals in China that have developed this technology. In order to prove that this technology has a significant effect on the treatment of cervical ossification of the posterior longitudinal ligament, we compared the efficacy of traditional ACCF surgery, in order to make the conclusion more true, we decided to carry out multi-center research.

Purpose: The aim of this study is to compare the effectiveness of clinical outcomes between ACAF surgery and Anterior cervical corpectomy decompression and fusion（ACCF）in patients with OPLL and CSS . A study hypothesis is that ACAF surgery outcomes will be equal even better and lower surgical complications which compared to ACCF surgery.

Methods: This study is a multi-center randomized clinical trial with randomized, controlled, multicenter research design. The OPLL patients will be randomly assigned in one of the two treatment groups: ACAF surgery and ACCF surgery. Five outcome measures will be collected pre-operative for baseline, and then at1, 12, 24, 48, 96,240weeks post-operative follow-up visits, including: (1)JOA) .(2)VAS. (3)NURIC Graded .(4)NDI . (5) radiological parameter. After randomization, the ACAF group will receive anterior controllable antedisplacement and fusion and the ACCF group will receive anterior cervical corpectomy decompression and fusion.

DETAILED DESCRIPTION:
Background: Although anterior and posterior decompression surgery are both reported to treat patients with myelopathy caused by OPLL（Posterior longitudinal ligament ossification）. The surgical strategy of the disease is still controversial when the OPLL is multilevel and severe. Novel techniques for better and safer results are required. Dr. Shi recently proposed a new technique as Ossification of anterior decompression surgery, which is also called anterior controllable antedisplacement and fusion (ACAF) , for ossification of the posterior longitudinal ligament (OPLL) with myelopathy. The ACAF technology has been in clinical trials for some time. More and more doctors are starting to pay attention to this technology. There are many hospitals in China that have developed this technology. In order to prove that this technology has a significant effect on the treatment of cervical ossification of the posterior longitudinal ligament, we compared the efficacy of traditional ACCF surgery, in order to make the conclusion more true, we decided to carry out multi-center research.

Purpose: The aim of this study is to compare the effectiveness and safety of clinical outcomes between ACAF surgery and Anterior cervical corpectomy decompression and fusion（ACCF）in patients with OPLL. A study hypothesis is that ACAF surgery outcomes will be equal even better and lower surgical complications which compared to ACCF surgery.

Methods: This study is a multi-center randomized clinical trial with randomized, controlled, multicenter research design. The OPLL patients will be randomly assigned in one of the two treatment groups: ACAF surgery and ACCF surgery. Five outcome measures will be collected pre-operative for baseline, and then at1, 12, 24, 48, 96,240weeks post-operative follow-up visits, including : (1) Japanese Orthopaedic Association (JOA) scales to assess the spinal cord functions.(2)Visual analogue scale (VAS) to assess pain relief. (3)NURIC Graded to assess walking function.(4) Neck Disabilitv Index(NDI) to assess cervical function . (5) radiological parameters to assess ossification forward distance. And the pre & postoperative radiological parameters, and surgical complications were also investigated. The investigator performing the outcome measures will be blinded to group assignment, and therefore will not participate in treatment. After randomization, the ACAF group will receive anterior controllable antedisplacement and fusion and the ACCF group will receive anterior cervical corpectomy decompression and fusion.

Data Analysis: T test or wilcoxon rank sum test will be used to examine the differences in the five measures between groups and at the six different time frames with the α level set at 0.05. Chi square test will be used to compare the differences in the surgical complications data over time and between groups.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 45-70 years, without gender limitation, are willing to sign informed consent;
2. patients diagnosed with posterior longitudinal ligament ossification of the cervical spine;
3. patients with limbs numbness, walking instability, banding and other spinal cord, nerve root compression symptoms, may be associated with urinary dysfunction, conservative treatment is invalid or gradually increased;

Exclusion Criteria:

1. Cervical ligamentous ossification, cervical trauma, cervical cancer, cervical tuberculosis and other inflammatory diseases;
2. accompanied by thoracolumbar spine and other spine parts of the disease affect the clinical symptoms of patients;
3. associated with amyotrophic lateral sclerosis and other motor neuron diseases and other neurological diseases;
4. poor health condition, unable to tolerate surgery;
5. patients (or their guardians) can not give full informed consent for adult dysfunction;
6. patients who have participated in other clinical trials in the past 1 month
7. patients with active hepatitis B (including HBeAg) or serological markers (HBsAg or / and HBeAg or / and HBcAb), hepatitis C, tuberculosis, cytomegalovirus infection, severe fungal infection or HIV infection;
8. patients with active peptic ulcers within 3 months before randomization;
9. patients with malignant neoplasms;
10. Vertebral length more than 3 intervertebral spaces.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes of patient-reported scores assessing improvement of spinal cord function underwent ACAF surgery compared to ACCF surgery | At 1 week pre- and 1, 12, 24, 48,96，240 weeks post-operative follow-up visits.
  JOA total score up to 17 points, the lowest 0 points. The lower the score, the more obvious the dysfunction. Improvement index = post-treatment score - pre-treatment score, post-treatment score improvement rate = [(post-treatment score - pre-treatment score) / 17 - pre-treatment score] × 100%. By improving the index can reflect the improvement of patients before and after treatment and clinical efficacy. The improvement rate can also correspond to the commonly used efficacy criteria: cure is 100% improvement, improvement is greater than 60% effective, 25-60% is effective, and less than 25% is ineffective.

SECONDARY OUTCOMES:
Changes of patient-reported scores assessing improvement of Walking function underwent ACAF surgery compared to ACCF surgery | At 1 week pre- and 1, 12, 24, 48,96，240 weeks post-operative follow-up visits.
  NURIC Graded presented by NURIC in 1972 used to assess improvement of Walking function。s divided into 6 levels, 0 - Although there are symptoms, but not based on the basis of spinal cord involvement (no limb numbness, decreased muscle strength and other symptoms); Grade 1 - spinal cord involvement (numbness of the limbs, decreased muscle strength and other symptoms), but normal gait; Level 2 ---- mild gait abnormalities, does not affect the work; Level 3 ---- abnormal gait, affecting work; Level 4 ---- Need to support before walking; Level 5 ---- can not walk.
Changes of patient-reported scores assessing improvement of pain underwent ACAF surgery compared to ACCF surgery | At 1 week pre- and 1, 12, 24, 48,96，240 weeks post-operative follow-up visits.
  Visual Analogue Scale/Score（VAS） score used to assess improvement of pain.This method is more sensitive and comparable. Draw a 10 cm horizontal line on the paper, one end of the horizontal line is 0, said no pain; the other end of 10, said the pain; the middle part of the pain of varying degrees.
Changes of patient-reported scores assessing improvement of quality of life and cervical function underwent ACAF surgery compared to ACCF surgery | At 1 week pre- and 1, 12, 24, 48,96，240 weeks post-operative follow-up visits.
  Neck Disabilitv Index（NDI) used to assess improvement of Quality of life and cervical function.Clinical assessment of cervical function is commonly used, the scale includes the degree of pain, personal food, carrying objects, reading, headache, attention, work, driving, sleep and entertainment in all aspects. Each 5 points, the total score from 0 points (barrier-free) to 50 points (completely paralyzed), the higher the score the heavier the dysfunction.
Changes of patient-reported scores assessing ossification and spinal cord forward distance underwent ACAF surgery compared to ACCF surgery | At 1 week pre- and 1, 12, 24, 48,96，240 weeks post-operative follow-up visits.
  radiological parameters used to assess assessing ossification and spinal cord forward distance.The results for the direct measurement of CT and MRI results, the minimum 0mm, the maximum 10mm, the greater the distance forward, indicating that the wider spinal canal, the better the spinal cord decompression, the better the surgical results.

CONTACTS AND LOCATIONS:
Overall Officials: Jiangang MI: Last Name:, Study Chair — Shanghai Changzheng Hospital, Second Military Medical University
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sun JC, Zhang B, Shi J, Sun KQ, Huan L, Sun XF, Liu N, Zheng B, Wang HB. Can K-Line Predict the Clinical Outcome of Anterior Controllable Antedisplacement and Fusion Surgery for Cervical Myelopathy Caused by Multisegmental Ossification of the Posterior Longitudinal Ligament? World Neurosurg. 2018 Aug;116:e118-e127. doi: 10.1016/j.wneu.2018.04.128. Epub 2018 Apr 27. PMID 29709746
- [Background] Yang H, Sun J, Shi J, Yang Y, Guo Y, Zheng B, Wang Y. In Situ Decompression to Spinal Cord During Anterior Controllable Antedisplacement Fusion Treating Degenerative Kyphosis with Stenosis: Surgical Outcomes and Analysis of C5 Nerve Palsy Based on 49 Patients. World Neurosurg. 2018 Jul;115:e501-e508. doi: 10.1016/j.wneu.2018.04.078. Epub 2018 Apr 22. PMID 29689396
- [Background] Yang H, Sun J, Shi J, Shi G, Guo Y, Yang Y. Anterior Controllable Antedisplacement Fusion (ACAF) for Severe Cervical Ossification of the Posterior Longitudinal Ligament: Comparison with Anterior Cervical Corpectomy with Fusion (ACCF). World Neurosurg. 2018 Jul;115:e428-e436. doi: 10.1016/j.wneu.2018.04.065. Epub 2018 Apr 17. PMID 29678703
- [Background] Miao J, Sun J, Shi J, Chen Y, Chen D. A Novel Anterior Revision Surgery for the Treatment of Cervical Ossification of Posterior Longitudinal Ligament: Case Report and Review of the Literature. World Neurosurg. 2018 May;113:212-216. doi: 10.1016/j.wneu.2018.02.076. Epub 2018 Feb 21. PMID 29476997
- [Background] Sun JC, Yang HS, Shi JG, Yuan W, Xu XM, Shi GD, Jia LS. Morphometric Analysis of the Uncinate Process as a Landmark for Anterior Controllable Antedisplacement and Fusion Surgery: A Study of Radiologic Anatomy. World Neurosurg. 2018 May;113:e101-e107. doi: 10.1016/j.wneu.2018.01.181. Epub 2018 Feb 5. PMID 29421454
- [Background] Sun J, Shi J, Xu X, Yang Y, Wang Y, Kong Q, Yang H, Guo Y, Han D, Jiang J, Shi G, Yuan W, Jia L. Anterior controllable antidisplacement and fusion surgery for the treatment of multilevel severe ossification of the posterior longitudinal ligament with myelopathy: preliminary clinical results of a novel technique. Eur Spine J. 2018 Jun;27(6):1469-1478. doi: 10.1007/s00586-017-5437-4. Epub 2017 Dec 28. PMID 29285560